CLINICAL TRIAL: NCT03647878
Title: Prospective Non-interventional Study of Cabozantinib as Monotherapy or in Combination With Nivolumab in Patients With Advanced or Metastatic Renal Cell Carcinoma Under Real-life Clinical Setting in 1st Line Treatment
Brief Title: Study of Cabozantinib as Monotherapy or in Combination With Nivolumab in Patients With Advanced or Metastatic Renal Cell Carcinoma Under Real-life Clinical Setting in 1st Line Treatment.
Acronym: CABOCARE
Status: Active, not recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-DE-60000-009
Record Dates: First submitted 2018-07-25; First posted 2018-08-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the protocol, is to describe the use of cabozantinib tablets as monotherapy or in combination with nivolumab including the number of dose reductions, dose interruptions and terminations due to (serious) adverse events in subjects with advanced or metastatic renal cell carcinoma (mRCC) treated in real-life clinical setting in 1st line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years and older with capacity to consent.
* Subjects receiving cabozantinib as monotherapy or in combination with nivolumab as a first line treatment for advanced or metastatic renal cell carcinoma
* Subjects with the intention to be treated with cabozantinib tablets as monotherapy or in combination with nivolumab according to the current local Summary of Product Characteristics (SmPC); decision has to be taken before entry in the study.
* Signed written informed consent

Exclusion Criteria:

* Participation in an interventional study at the same time and/or within 3 months before baseline.
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Cabozantinib as monotherapy or in combination with nivolumab in advanced or metastatic renal cell carcinoma in 1st line treatment
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with dose reduction of cabozantinib due to Serious Adverse Events/Adverse Events (SAEs/AEs) | 2 years
  The proportion of subjects with ≥1 dose reduction due to AE will be described with its 95% confidence interval, by risk group and overall.
The proportion of subjects with dose interruption of cabozantinib and/or nivolumab due to SAEs/AEs | 2 years
  The proportion of subjects with ≥1 dose interruption due to AE will be described with its 95% confidence interval, by risk group and overall.
The proportion of subjects with termination of cabozantinib /cabozantinib-nivolumab combination due to SAEs/AEs | 2 years
  The proportion of subjects with ≥1 discontinuation due to AE will be described with its 95% confidence interval, by risk group and overall.
Number of injection delayed of nivolumab due to SAE/AE | 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival is defined as the time between the start date of cabozantinib and the date of progression or death from any cause. Disease progression is defined as either radiological progression assessed by the investigator using RECIST 1.1 or clinical progression.
Best overall response - Overall Response Rate (ORR) | 2 years
  The best overall response is the best response assessed by investigator recorded during the treatment period. ORR is defined as the proportion of subjects achieving complete or partial response.
Best overall response - Disease Control Rate (DCR) | 2 years
  The best overall response is the best response assessed by investigator recorded during the treatment period. DCR is defined as the proportion of subjects achieving a complete response, partial response or stable disease.
All non-serious and serious adverse events (AEs / SAEs) and fatal outcomes | 2 years
  Safety: clinical parameter, as routinely assessed by the investigator, as well as occurrence of all serious and non-serious AEs as well as fatal outcomes and special situations. The adverse events will be described overall and also according to level of physical activity assessed by questionnaire and actigraph.
Impact of the activity level at baseline on the occurrence of adverse events (AEs) | 2 years
  Safety: clinical parameter, as routinely assessed by the investigator, as well as occurrence of all serious and non-serious AEs as well as fatal outcomes and special situations; data of activity level and quality of life will be collected using the quality of life questionnaire (NFKSI-19 questionnaire) and the activity questionnaire; inflammatory blood markers, as routinely assessed by the investigator, will be captured.
The proportion of subjects with termination due to SAEs/AEs in sub-group | 2 year
  The proportion of subjects with ≥1 termination due to AE will be described with its 95% confidence interval, by risk group and overall split by histological subtype (clear cell and non-clear cell).
The proportion of subjects with dose interruption due to SAEs/AEs in sub-group | 2 year
  The proportion of subjects with ≥1 dose interruption due to AE will be described with its 95% confidence interval, by risk group and overall split by histological subtype (clear cell and non-clear cell).
The proportion of subjects with dose reduction due to SAEs/AEs in sub-group | 2 years
  The proportion of subjects with ≥1 dose reduction due to AE will be described with its 95% confidence interval, by risk group and overall split by histological subtype (clear cell and non-clear cell).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (82):
- Austria (5):
  - Landeskrankenhaus Hochsteiermark, Leoben
  - Kepler Universitätsklinikum GmbH, Linz
  - Uniklinikum Salzburg, Salzburg
  - Salzkammergutklinikum Vöcklabruck, Vöcklabruck
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Germany (77):
  - Universitätsklinikum Aachen, Aachen
  - Urologisches Zentrum Euregio, Aachen
  - Onkologie aschaffenburg, Aschaffenburg
  - Universitätsklinikum Augsburg A.ö.R, Augsburg
  - MVZ Taunus GmbH, Bad Homburg
  - Hämatologisch-Onkologische Schwerpunktpraxis, Bad Liebenwerda
  - Urologische Praxis Bad Schlema, Bad Schlema
  - Klinikum am Bruderwald Medizinische Klinik V, Bamberg
  - GFO Kliniken Rhein-Berg, Bergisch Gladbach
  - Praxis für Urologie, Berlin
  - Onkologie am Segelfliegerdamm, Berlin
  - Praxis am Volkspark, Berlin
  - Praxis Urologie Köpenick, Berlin
  - Urologische Praxis Berlin, Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Zentrum für urologische Onkologie, Palliativmedizin und allgemeine Urologie, Berlin
  - Urologische Arztpraxis, Bernburg
  - Franziskus Hospital Bielefeld, Bielefeld
  - Centrum für Operative Urologie, Bremen
  - Klinikum Bremen Mitte, Bremen
  - Edia.med MVZ, Chemnitz
  - Gemeinschaftspraxis für Urologie Cottbus, Cottbus
  - Onkologisches Zentrum Donauwörth, Donauwörth
  - Onkozentrum Dresden/Freiberg, Dresden
  - Urologische Gemeinschaftspraxis, Dresden
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden, Dresden
  - Fachzentrum für Urologie Eggenfelden, Eggenfelden
  - St. Georg Klinikum, Eisenach
  - Urologische Arztpraxis, Eisleben Lutherstadt
  - Uniklinikum Erlangen, Erlangen
  - Markuskrankenhaus, Frankfurt am Main
  - Gemeinschaftspraxis, Garbsen
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Göttingen, Göttingen
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Asklepios Klinik Altona, Hamburg
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Onkologisches Studienzentrum am Raschplatz, Hanover
  - Immunologisch onkologisches MVZ, Hanover
  - Kreiskliniken Herford, Herford
  - Uniklinik Jena, Jena
  - Praxis für Hämatologie, Onkologie und Gerinnung, Kronach
  - Onkologische Schwerpunktpraxis, Kronach
  - Studienzentrum UnterEms, Leer
  - Urologische Arztpraxis, Leipzig
  - Urologische Praxis, Luckenwalde
  - Universitätsklinikum Magdeburg, Magdeburg
  - Uniklinik Marburg, Marburg
  - Praxis für Urologie, Andrologie, Onkologie und medikamentöse Tumortherapie, Markkleeberg
  - Onkologische Praxis Moers, Moers
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Facharztpraxis für Hämatologie und Internistische Onkologie, München
  - LMU Urologische Klinik und Poliklinik, München
  - Universitätsklinikum Münster, Münster
  - Praxis Naunhof, Naunhof
  - Urologische Gemeinschaftspraxis, Neunkirchen
  - Praxis für Hämatologie und Internistische Onkologie, Neustadt am Rübenberge
  - Klinikum Nürnberg, Nuremberg
  - MVZ Urologie gGmbH, Nuremberg
  - Sana Klinikum Offenbach GmbH, Offenbach
  - MVZ Kreis Olpe, Olpe
  - Klinikum Osnabrück GmbH, Osnabrück
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Urologische Praxis, Parchim
  - Urologie, Potsdam
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Elblandklinikum Riesa, Riesa
  - MVZ MP Saaletal, Saalfeld
  - Zentrum für Ambulante Onkologie, Schorndorf
  - Klinikum Sindelfingen-Böblingen, Sindelfingen
  - Klinikum Solingen, Solingen
  - Krankenhaus Torgau J. Kentmann gGmbH, Torgau
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Medizinische Studiengesellschaft Nord-West GmbH, Westerstede
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - GIM - Gemeinschaftspraxis Innere Medizin, Witten
  - Praxis Urologie Köpenick, Zwickau

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/